CLINICAL TRIAL: NCT00454428
Title: Randomized Trial of Pulsatile vs Non Pulsatile Perfusion on Short Term Changes in Kidney Function Using an Intra-Aortic Ballooon Pump During Cardioplegic Arrest in Patients Undergoing Myocardial Reperfusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Catanzaro (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 27579
Record Dates: First submitted 2007-03-29; First posted 2007-03-30 (Estimated); Last update posted 2007-03-30 (Estimated); Status verified 2006-03

CONDITIONS: Aortocoronary Bypass
Keywords: Bypass Surgery; Coronary Artery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: pulsatile intra-aortic balloon pump

SUMMARY:
Linear flow during cardiopulmonary bypass (CPB) frequently induces renal damage.

We will evaluate whether automatic intra-aortic balloon pump (IABP) induce pulsatile perfusion preserves renal function in patients undergoing myocardial revascularization at different risk for renal damage.

100 patients undergoing preoperative IABP will be stratified for renal function.

Intervention. The patients will be randomized to non-pulsatile CPB during cardioplegic arrest or automatic IABP induced pulsatile CPB.

Renal function, daily diuretics, complication rate, lactatemia and other biochemical indices will be compared in patients.

We will prospectively enrolle 100 patients undergoing isolated primary high-risk coronary artery bypass grafting for severe left main stem disease (70% narrowing) or left-main equivalent three-vessels coronary disease. On admission to our institution, the patients will be stratified for renal function according to KDOQI and randomly assigned to Group A or Group B. We will exclude from the study patients older than 75 years, and/or with kidney disease ≥ Stage 4 (GFR 15 - 29 ml/min/1.73 m2), and/or with other splanchnic organ comorbidities (liver or mesenteric impairment, abdominal aortic aneurysm, abdominal arteries vasculopathy), and/or severe autoimmune disease.

The patients randomized to Group A (n=50) will receive a preoperative IABP treatment before induction of anesthesia, with IABP turned off during cardioplegic arrest, and restarted with a 1:1 IABP mode immediately after cross-clamp removal (as is the traditionally adopted perioperative IABP support); the other 50 (Group B) will receive standard preoperative treatment with IABP, which will switche into an automatic 80 bpm mode during cross-clamp time, and switche again into a 1:1 IABP after cross-clamp removal, in order to achieve a pulsatile perfusion during the entire intra-operative time-course.

The patients will be stratified in 2 subgroups according to the preoperative renal function: a subgroup will include 64 patients (32 allocated in Group A and 32 in Group B) with stage 1 or 2 [Stage 1: GFR ≥90 ml/min/1.73 m2 - Stage 2: GFR 60 - 89 ml/min/1.73 m2] and therefore considered at lower-risk for post-CPB renal damage; the remaining 36 (18 for each group) with KDOQI Stage 3 of kidney disease (GFR 30 - 59 ml/min/1.73 m2) will be considered at higher-risk for perioperative renal complications [19].

DETAILED DESCRIPTION:
Linear flow during cardiopulmonary bypass (CPB) frequently induces renal damage.

We will evaluate whether automatic intra-aortic balloon pump (IABP) induced pulsatile perfusion preserves renal function in patients undergoing myocardial revascularization at different risk for renal damage.

100 patients undergoing preoperative IABP will be stratified for renal function.

Intervention. The patients will be randomized to non-pulsatile CPB during cardioplegic arrest or automatic IABP induced pulsatile CPB.

Renal function, daily diuretics, complication rate, lactatemia and other biochemical indices will be compared in patients.

We will prospectively enrolle 100 patients undergoing isolated primary high-risk coronary artery bypass grafting for severe left main stem disease (70% narrowing) or left-main equivalent three-vessels coronary disease. On admission to our institution, the patients will be stratified for renal function according to KDOQI and randomly assigned to Group A or Group B. We will exclude from the study patients older than 75 years, and/or with kidney disease ≥ Stage 4 (GFR 15 - 29 ml/min/1.73 m2), and/or with other splanchnic organ comorbidities (liver or mesenteric impairment, abdominal aortic aneurysm, abdominal arteries vasculopathy), and/or severe autoimmune disease.

The patients randomized to Group A (n=50) will receive a preoperative IABP treatment before induction of anesthesia, with IABP turned off during cardioplegic arrest, and restarted with a 1:1 IABP mode immediately after cross-clamp removal (as is the traditionally adopted perioperative IABP support); the other 50 (Group B) will receive standard preoperative treatment with IABP, which will switche into an automatic 80 bpm mode during cross-clamp time, and switche again into a 1:1 IABP after cross-clamp removal, in order to achieve a pulsatile perfusion during the entire intra-operative time-course.

The patients will be stratified in 2 subgroups according to the preoperative renal function: a subgroup will include 64 patients (32 allocated in Group A and 32 in Group B) with stage 1 or 2 [Stage 1: GFR ≥90 ml/min/1.73 m2 - Stage 2: GFR 60 - 89 ml/min/1.73 m2] and therefore considere at lower-risk for post-CPB renal damage; the remaining 36 (18 for each group) with KDOQI Stage 3 of kidney disease (GFR 30 - 59 ml/min/1.73 m2) will be considered at higher-risk for perioperative renal complications [19].

The study protocol has been approved by the institution's Ethical Committee/Institutional Review Board, and informed consent will be obtained from each patient.

Anesthesia Anesthetic technique will be standardized: induction will consiste of i.v. propofol infusion (3 mg/kg) combined with fentanyl (0.10 mg/Kg). Neuromuscular blockade will be achieved by 4 mg/h pancuronium bromide, and lungs will be ventilated to normocapnia with air and oxygen (45-50%). Propofol infusion (150-200 μg/Kg per min) and isoflurane (0.5% inspired concentration) will maintaine anesthesia. Inotropes will be started immediately after aortic cross-clamp removal to maintain adequate mean systemic pressure, always starting with enoximone at a dosage of 5 μg/Kg/min. The need for further increase in inotropes will be record: inotropes will be defined as "low-dose" when enoximone will be administered at a dosage 5 μg/Kg/min, "medium-dose" when enoximone will be between 6 and 10 μg/Kg/min, or dobutamine will add at a dosage between 5 and 10 μg/Kg/min, and "high-dose" when enoximone or dobutamine will be >10 μg/Kg/min or epinephrine add at any dose.

Surgical technique and cardiopulmonary bypass According to our Institutional policy we will insert IABP (7.5 or 8 Fr, 34 or 40 ml according to the body surface area; balloon Datascope Corp., Fairfield, NJ, connected to a Datascope pump [Datascope Corp, Fairfield, NJ]) percutaneously with the "sheetless" technique, through the best femoral artery, before induction of anesthesia, in order to better support the perioperative hemodynamic of patients undergoing surgery for severe left main stem or 3-vessels left-main equivalent disease. The correct placement of IABP will be always assessed by postoperative chest X-ray or transesophageal echocardiography. Patients will receive anticoagulation with enoxaparin, with a target activated partial thromboplastin time >40 seconds, starting when the postoperative bleeding was controlled (usually within 6 hours). IABP will be withdrawn when hemodynamic stability will restore (i.e., a cardiac index 2.0 L/m2 per minute with only minimal pharmacologic inotropic support, dobutamine or enoximone at 5 µg/kg per minute). CPB and surgical techniques will be standardized and not changed during the study period. Heparin will be given at a dose of 300 IU/kg to achieve a target activated clotting time of 480 seconds or above. Blood recovery with an autotransfusion device (Autotrans Dideco, Mirandola, Modena, Italy) will be performed intraoperatively in all cases. A level of hemoglobin lower than 8 g/dl will be used as an indication for blood transfusion. Standard CPB circuit will be used. The extracorporeal circuit will be primed with 1000 ml of Ringer's Lactate solution and 40 mg of heparin. Systemic temperature will be kept between 32 and 34° C. Myocardial protection will be achieved with intermittent antegrade and retrograde hyperkalemic blood cardioplegia. Total CPB flow will be maintained at 2.6 L/min-1/m-2. In Group A patients, IABP will be turned off during cardioplegic arrest, maintaining a standard non-pulsatile CPB; Group B patients will undergo IABP-induced pulsatile CPB during cardioplegic arrest, with pulsatile flow maintained by an automatic 80 bpm mode until aortic declamping.

Endpoints The primary endpoint of this study is the evaluation of the renal function as assessed by measuring GFR in the perioperative period. In all patients will be evaluated perioperative renal function, in-hospital mortality and morbidity, and complications, in-hospital and intensive therapy unit (ITU) stay, IABP-related complications. Renal function is primarily evaluated by GFR calculated using the abbreviated Modification of Diet in Renal Disease (MDRD) study equation, recommended by KDOQI as the preferred equation for the calculation of GFR in adults (taking into account serum creatinine, age, race, gender) [22] and, secondarily, by other indices, such as urine output, need for diuretics, blood urea nitrogen (BUN). Plasma lactate concentrations will be measured to indirectly assess the adequacy of tissue perfusion [20] Acute renal insufficiency (ARI) is defined as a decrease greater than 50% over preoperative value of calculated GFR. Acute renal failure (ARF) is defined as any postoperative renal insufficiency requiring first-time hemofiltration, dialysis or any other renal replacement therapy (RRT). In-hospital mortality is defined as any death occurring during hospital stay or in the first 30 postoperative days. Hospital morbidity is defined as any complication requiring specific therapy or causing a delay in hospital or ITU discharge. IABP-related complications is defined as any aortic dissection or perforation, limb or mesenteric ischemia, or infection or hemorrhage at the balloon entry point.

Biochemical analysis All patients will undergo pre- and perioperatively routine laboratory investigations, including standard hemogram, serum levels of creatinine, urea nitrogen, calcium, phosphate, glucose, albumin, electrolytes, albumin, transaminases, -glutamyl-transpeptidase, lactic acid dehydrogenase, bilirubin, acid-base parameters, troponin I and lactic acid. The determinations of the majority of these parameters will be conducted preoperatively before anesthetic induction, and at 12, 24, 48, and 72 hours postoperatively. In order to evaluate the adequacy of myocardial protection techniques, Troponin I will be measured on coronary sinus blood samples, obtained from the retrograde cardioplegic cannula, 10 minutes following completion of proximal anastomoses. The Troponin I assays will be carried out using diagnostic kits provided by Beckman Coulter (Fullerton, California; AccuTnITM Access Immunoassay System).

Statistical analysis Statistical analysis will be performed by the SPSS program for Windows, version 10.1 (SPSS Inc, Chicago, IL). Continuous variables will be presented as mean ± standard deviation, and categorical variables as absolute numbers and/or percentages. Data will be checked for normality before statistical analysis. Normally-distributed continuous variables will be compared using the unpaired t test, whereas the Mann-Whitney U test will be used for those variables that are not normally distributed. Categorical variables will be analyzed using either the chi-square test or Fischer's exact test. Comparison between and within groups will be made using two-way analysis of variance for repeated measures. Comparisons will be considered significant if p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing isolated primary high-risk coronary artery bypass grafting for severe left main stem disease (70% narrowing) or left-main equivalent three-vessels coronary disease

Exclusion Criteria:

* Patients older than 75 years
* With kidney disease ≥ Stage 4 (GFR 15 - 29 ml/min/1.73 m2)
* With other splanchnic organ comorbidities (liver or mesenteric impairment, abdominal aortic aneurysm, abdominal arteries vasculopathy)
* Severe autoimmune disease.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Onorati, MD, Principal Investigator — cardiac surgery
Locations (1):
- Cardiac Surgery and Nephrology, Catanzaro, Catanzaro, Italy

REFERENCES:
- [Derived] Onorati F, Presta P, Fuiano G, Mastroroberto P, Comi N, Pezzo F, Tozzo C, Renzulli A. A randomized trial of pulsatile perfusion using an intra-aortic balloon pump versus nonpulsatile perfusion on short-term changes in kidney function during cardiopulmonary bypass during myocardial reperfusion. Am J Kidney Dis. 2007 Aug;50(2):229-38. doi: 10.1053/j.ajkd.2007.05.017. PMID 17660024